CLINICAL TRIAL: NCT03463317
Title: Left Atrial Appendage CLOSURE in Patients With Atrial Fibrillation at High Risk of Stroke and Bleeding Compared to Medical Therapy: a Prospective Randomized Clinical Trial
Brief Title: Left Atrial Appendage CLOSURE in Patients With Atrial Fibrillation Compared to Medical Therapy
Acronym: CLOSURE-AF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); Atrial Fibrillation Network (Other); Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Principal Investigator, Ulf Landmesser, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CLOSURE-AF-DZHK16
Record Dates: First submitted 2018-02-16; First posted 2018-03-13 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Anticoagulation; Left atrial appendage closure; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Aspirin; Clopidogrel; Dabigatran; Rivaroxaban; apixaban; edoxaban; Phenprocoumon; Warfarin

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, event-driven, randomized controlled trial (Following 2nd blinded interim analysis: no longer event-driven).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAA closure group (Experimental): Left atrial appendage closure by use of CE-mark approved LAA closure devices followed by post procedure treatment (antiplatelet therapy e.g. acetylsalicylic acid, clopidogrel)
  Interventions: Device: CE-mark approved LAA closure devices; Drug: Acetylsalicylic acid; Drug: Clopidogrel
- Best medical care group (Active Comparator): No left atrial appendage closure. Treatment with best medical care (NOACs (dabigatran, rivaroxaban, apixaban, edoxaban) or VKA (phenprocoumon, warfarin)
  Interventions: Drug: Dabigatran; Drug: Rivaroxaban; Drug: Apixaban; Drug: Edoxaban; Drug: Phenprocoumon; Drug: Warfarin

INTERVENTIONS:
Device: CE-mark approved LAA closure devices — LAA closure with post procedure treatment
  Arms: LAA closure group
Drug: Acetylsalicylic acid — post procedure treatment according to the physicians (recommendation are made in the protocol); oral anticoagulation is not prescribed in this group
  Other Names: ASS
  Arms: LAA closure group
Drug: Clopidogrel — post procedure treatment according to the physicians (recommendation are made in the protocol); oral anticoagulation is not prescribed in this group
  Arms: LAA closure group
Drug: Dabigatran — Patients allocated to the best medical care group receive either NOAC therapy or VKA
  Other Names: Pradaxa®
  Arms: Best medical care group
Drug: Rivaroxaban — Patients allocated to the best medical care group receive either NOAC therapy or VKA
  Other Names: Xarelto®
  Arms: Best medical care group
Drug: Apixaban — Patients allocated to the best medical care group receive either NOAC therapy or VKA
  Other Names: Eliquis®
  Arms: Best medical care group
Drug: Edoxaban — Patients allocated to the best medical care group receive either NOAC therapy or VKA
  Other Names: LIXIANA®
  Arms: Best medical care group
Drug: Phenprocoumon — Patients allocated to the best medical care group receive either NOAC therapy or VKA
  Other Names: Marcumar®
  Arms: Best medical care group
Drug: Warfarin — Patients allocated to the best medical care group receive either NOAC therapy or VKA
  Other Names: Coumadin®
  Arms: Best medical care group

SUMMARY:
The study goal is to determine the clinical benefit of percutaneous catheter-based left atrial appendage (LAA) closure in patients with non-valvular atrial fibrillation (NVAF) at high risk of stroke (CHA2DS2-VASc Score ≥2) as well as high risk of bleeding as compared to best medical care (including a [non-vitamin K] oral anticoagulant [(N)OAC] when eligible).

DETAILED DESCRIPTION:
The individualized therapy with oral anticoagulants is considered to be an essential preventive therapy in patients with atrial fibrillation. The risk of stroke can be reduced by approximately 65%. However, long-term anticoagulation therapy also increases the risk of major bleeding.

A significant proportion of patients at high risk of stroke do not tolerate long-term anticoagulation due to various relative or absolute contraindications. As demonstrated in previous studies with non-vitamin K antagonist anticoagulants (NOAK), 20-25% of patients were unable to tolerate long-term anticoagulation therapy.

For this reason, additional therapeutic approaches for stroke prevention in patients with atrial fibrillation have been developed.

A promising approach is catheter-based closure of the left atrial appendage, because more than 90% of cardiac thrombi in patients with non-valvular atrial fibrillation are detected in the left atrial appendage. Recent registry studies show that the safety of LAA occluder implantation is promising. However, further scientific studies are required, in order to explore more benefits of the underlying method and eligible patients for implantation.

Study objectives:

The study goal is to determine the clinical benefit of percutaneous catheter-based left atrial appendage (LAA) closure in patients with non-valvular atrial fibrillation (NVAF) at high risk of stroke (CHA2DS2-VASc Score ≥2) as well as high risk of bleeding as compared to best medical care (including a [non-vitamin K] oral anticoagulant [(N)OAC] when eligible).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Documented atrial fibrillation (paroxysmal, persistent, long-standing persistent or permanent)
* CHA2DS2VASc-Score ≥2
* High risk of bleeding under oral anticoagulation or contraindication for (N)OAC therapy, in particular patients with at least one of the following conditions:

  * HAS-BLED-Score ≥3
  * Prior intracranial/intraspinal bleed, intraocular bleed compromising vision (BARC: type 3c)
  * Hemorrhagic/bleeding complication fulfilling BARC type 3a or 3b: gastrointestinal tract, genitourinary tract or respiratory tract bleeding, where the patient is considered to be at a persistently increased risk of bleeding, e.g. the cause of bleeding cannot be successfully eliminated
  * Chronic kidney disease with eGFR 15-29 ml/min/1.73 m2
  * Any recurrent bleeding making chronic anticoagulation not feasible
* Subject eligible for an LAA occluder device
* Age ≥18 years
* Willing and capable of providing informed consent, participating in all associated study activities
* negative SARS-CoV-2 PCR test (no longer than 48 hours prior to randomization in outpatients or not older than 14 days in continuously hospitalized patients without signs of COVID-19 infection) or negative SARS- CoV-2 rapid antigen test (no longer than 24 hours prior to randomization)

Exclusion Criteria:

* Absolute contraindication to acetylsalicylic acid
* Comorbidities other than AF requiring chronic (N)OAC therapy, e.g. mechanical heart valve prosthesis
* Symptomatic carotid disease (if not treated)
* Complex aortic atheroma with mobile plaque (Kronzon classification grade V)
* Heart transplant
* Active infection or symptoms suggestive of COVID-19 infection or active endocarditis or other infections resulting in bacteremia
* Cardiac tumor
* Severe liver failure (Child-Pugh class C or liver failure with coagulopathy)
* Severe renal failure (GFR <15 ml/min/1.73m2 or current requirement for dialysis defined as current, regular renal replacement therapy performed at least weekly including hemodialysis and peritoneal dialysis within the last 30 days)
* Pregnancy or breastfeeding
* For female patients of reproductive potential: Unwilling to agree to use a highly effective method of contraception (Pearl index <1) throughout the study period
* Subject with participation in another interventional clinical trial during this study or within 30 days before entry into this trial.
* Known terminating disease with life expectancy <1 year (including those with end-stage heart failure)
* Subjects, who are committed to an institution due to binding official or court order
* Subject who is dependent on the Site, the Site Investigator, any sub- investigator, his/her representative and/or the sponsor
* Persons who are not proficient in the German language
* Unstable/not fully recompensated acute heart failure corresponding to NYHA class III and/or IV
* Subjects with known antiphospholipid syndrome
* Subjects with planned cardiac or non-cardiac surgery or intervention. (These subject can be included 30 days after such intervention / surgery.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 912 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Primary endpoint (net clinical benefit) | After 3, 6, and 12 months. Twice a year until 24 months and once a year after 24 months.
  Survival time free of the composite of:
  * Stroke (including ischemic or hemorrhagic stroke)
  * Systemic embolism
  * Major bleeding (BARC type 3-5)
  * Cardiovascular or unexplained death

SECONDARY OUTCOMES:
Primary endpoint events per year | After 3, 6, and 12 months. Twice a year until 24 months and once a year after 24 months.
  assessed by the number of primary endpoint events during the follow-up period.
Combined endpoint: MACCE | After 3, 6, and 12 months. Twice a year until 24 months and once a year after 24 months.
  (stroke/systemic embolism/cardiovascular death/myocardial infarction)
Mortality | After 3, 6, and 12 months. Twice a year until 24 months and once a year after 24 months.
  (including all-cause death, cardiovascular death, non- cardiovascular death, peri-procedural death)
Major bleeding | After 3, 6, and 12 months. Twice a year until 24 months and once a year after 24 months.
  BARC type 3-5 (according to the BARC (Bleeding Academic Research Consortium) definition for bleeding).
Systemic embolism | After 3, 6, and 12 months. Twice a year until 24 months and once a year after 24 months.
  assessed by the rate of systemic embolism during the follow-up period.
Ischemic stroke | After 3, 6, and 12 months. Twice a year until 24 months and once a year after 24 months.
  Stroke will be assessed according to 2014 ACC/AHA Key Data Elements and Definitions for Cardiovascular Endpoint Events in Clinical Trials: A Report of the American College of Cardiology/AmericanHeart Association Task Force on Clinical Data Standards (Writing Committee to Develop Cardiovascular Endpoints Data Standards). J Am Coll Cardiol, 2015.
Hemorrhagic stroke | After 3, 6, and 12 months. Twice a year until 24 months and once a year after 24 months.
  Stroke will be assessed according to 2014 ACC/AHA Key Data Elements and Definitions for Cardiovascular Endpoint Events in Clinical Trials: A Report of the American College of Cardiology/AmericanHeart Association Task Force on Clinical Data Standards (Writing Committee to Develop Cardiovascular Endpoints Data Standards). J Am Coll Cardiol, 2015.
Transient ischemic attack | After 3, 6, and 12 months. Twice a year until 24 months and once a year after 24 months.
  Defined as neurological deficit of vascular origin lasting ≤24 hours without corresponding brain lesion. TIA will be assessed according to 2014 ACC/AHA Key Data Elements and Definitions for Cardiovascular Endpoint Events in Clinical Trials: A Report of the American College of Cardiology/AmericanHeart Association Task Force on Clinical Data Standards (Writing Committee to Develop Cardiovascular Endpoints Data Standards). J Am Coll Cardiol, 2015.
Myocardial infarction | After 3, 6, and 12 months. Twice a year until 24 months and once a year after 24 months.
  Myocardial infarction will be assessed according to the third universal definition of myocardial infarction (Eur Heart J, 2012).
Hospitalization for bleeding or cardiovascular event | After 3, 6, and 12 months. Twice a year until 24 months and once a year after 24 months.
  Hospitalization for bleeding or cardiovascular event will be assessed according to 2014 ACC/AHA Key Data Elements and Definitions for Cardiovascular Endpoint Events in Clinical Trials: A Report of the American College of Cardiology/AmericanHeart Association Task Force on Clinical Data Standards (Writing Committee to Develop Cardiovascular Endpoints Data Standards). J Am Coll Cardiol, 2015.
Changes in cognitive function | At day 0 and after 24 months.
  assessed by MoCA (= Montreal Cognitive Assessment). The MoCA will be used to assess the cognition of patients. Minimum score: 0 points, maximum score: 30 points.
Changes in health-related quality of life | At day 0 and after 6, and 12 months, twice a year until 24 months and once a year after 24 months of follow-up.
  assessed by EQ-5D-5L (German Version 1.0). The EQ-5D-5L consists of a 5-question multi-attribute questionnaire and a visual analogue self-rating scale. Minimum score: 0, maximum score: 100.
Changes in modified Ranking Scale (mRS) | At day 0, 1 day after implantation (device group only) and after 3, 12 and 24 months.

OTHER OUTCOMES:
Device-related complications | Until day 7 or discharge and after 3, 6,12 and 24 months.
  Device thrombus/fracture/erosion/infection/embolization, Pericardial effusion.
Procedure related death | Until day 7 or discharge and after 3, 6,12 and 24 months.
Technical and procedural success of device implantation | Until day 7 or discharge and after 3, 6,12 and 24 months.
Peri-procedural outcomes | At 7 days or discharge, 30 calendar days after implantation and after 3, 6,12 and 24 months.
Additionally, the total number of SAEs will be analyzed. | After 3, 6, and 12 months. Twice a year until 24 months and once a year after 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Landmesser, MD, Study Chair — Charite University, Berlin, Germany
Locations (42):
- Germany (42):
  - Charité Universitätsmedizin Berlin, Klinik für Kardiologie, Angiologie und Intensivmedizin, Deutsches Herzzentrum der Charité, Campus Benjamin Franklin (CBF), Berlin
  - DRK-Kliniken Berlin Köpenick, Klinik für Innere Medizin - Schwerpunkt Kardiologie und Angiologie, Berlin
  - Deutsches Herzzentrum der Charité, Klinik für Kardiologie, Angiologie und Intensivmedizin, Campus Virchow-Klinikum, Berlin
  - Klinik für Kardiologie, Angiologie und Intensivmedizin, Deutsches Herzzentrum der Charité, Campus Virchow-Klinikum (CVK), Berlin
  - Charité Universitätsmedizin Berlin, Campus Charité Mitte, Med. Klinik für Kardiologie und Angiologie, Berlin
  - Klinikum Brandenburg GmbH, Zentrum für Innere Medizin I, Brandenburg
  - Gesundheit Nord gGmbH, Klinikum Links der Weser, Klinik für Kardiologie und Angiologie, Bremen
  - Klinikum Coburg GmbH II. Med. Klinik für Innere Medizin und Kardiologie, Coburg
  - Amper Kliniken AG, Helios Amper-Klinikum Dachau, Innere Medizin I - Kardiologie & Pneumologie, Dachau
  - Städtisches Klinikum Dresden, II. Medizinische Klinik, Dresden
  - Technische Universität Dresden, Herzzentrum Dresden, Universitätsklinik, Medizinische Klinik Kardiologie, Dresden
  - Katholisches Krankenhaus "St. Johann Nepomuk", Klinik für Innere Medizin II - Kardiologie, Erfurt
  - HELIOS Klinikum Erfurt GmbH, 3. Medizinische Klinik, Erfurt
  - Universitätsklinikum Frankfurt, Medizinische Klinik III/ Kardiologie, Frankfurt
  - UHZ Freiburg Bad Krozingen Klinik für Kardiologie und Angiologie II, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Klinik für Kardiologie und Pneumologie, Göttingen
  - Universität Greifswald, Klinik für Innere Medizin B - Kardiologie, Greifswald
  - Universitätsklinikum Halle (Saale), Universitätsklinik und Poliklinik für Innere Medizin III, Halle
  - Asklepios Klinik Barmbek, I. Med. Abteilung - Kardiologie, Hamburg
  - Asklepios Klinik St. Georg Hamburg, Abteilung für Kardiologie, Hamburg
  - Cardiologicum Hamburg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Universitäres Herzzentrum, Klinik für Allgemeine und Interventionelle Kardiologie, Hamburg
  - Westküstenklinikum Heide Medizinische Klinik 2 - Kardiologie, Heide
  - Universitätsklinikum Heidelberg, Medizinische Klinik für Kardiologie, Angiologie und Pneumologie, Heidelberg
  - Oberhavel Kliniken, Klinik Hennigsdorf, Innere Medizin, Hennigsdorf
  - Universitätsklinikum Jena, Klinik für Innere Medizin I - Kardiologie, Jena
  - UKSH - Campus Kiel, Medizinische Klinik III - Kardiologie, Angiologie, Intensivmedizin, Kiel
  - Herzzentrum Leipzig, Universitätsklinik für Kardiologie, Leipzig
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Kardiologie, Leipzig
  - UKSH - Universitäres Herzzentrum Lübeck, Medizinische Klinik II - Kardiologie, Angiologie, Intensivmedizin, Lübeck
  - Universitätsmedizin Mainz, Kardiologie I - Zentrum für Kardiologie, Mainz
  - Universitätsmedizin Mannheim, I. Medizinische Klinik - Kardiologie, Angiologie, Intensivmedizin, Mannheim
  - Deutsches Herzzentrum München, Klinik an der TU München, München
  - LMU Universität München, Medizinische Klinik und Poliklinik I, München
  - Peter Osypka Herzzentrum München, München
  - Städt. Klinikum München GmbH, Klinikum Neuperlach, Klinik für Kardiologie, Pneumologie, intern. Intensivmedizin, München
  - Klinikum rechts der Isar, TU München, Klinik und Poliklinik für Innere Medizin I - Kardiologie, München
  - Universitätsmedizin Rostock, Herzzentrum, Zentrum Innere Medizin - Abteilung für Kardiologie, Rostock
  - Universitätsklinikum Tübingen, Medizinische Klinik, Abteilung III Kardiologie und Kreislauferkrankungen, Tübingen
  - Universitätsklinik Ulm, Klinik für Innere Medizin II - Kardiologie, Ulm
  - Universitätsklinikum Würzburg, Medizinische Klinik und Poliklinik I, Würzburg
  - Heinrich-Braun-Klinikum Zwickau, Klinik für Innere Medizin I - Kardiologie, Angiologie, Intern. Internsivmedizin, Zwickau

REFERENCES:
- [Derived] Landmesser U, Skurk C, Kirchhof P, Lewalter T, Hartung J, Rroku A, Pieske B, Brachmann J, Akin I, Jacobshagen C, Meder B, Zeiher A, Anker SD, Thiele H, Blankenberg S, Massberg S, Schunkert H, Frey N, Joost A, Bergmann M, Haeusler KG, Endres M, Wegscheider K, Boldt LH, Eitel I. Catheter-based left atrial appendage CLOSURE in patients with atrial fibrillation at high risk of stroke and bleeding as compared to best medical therapy: Rationale and design of the prospective randomized CLOSURE-AF trial. Am Heart J. 2026 Feb;292:107273. doi: 10.1016/j.ahj.2025.09.005. Epub 2025 Sep 12. PMID 40946883
- See also: trial website — https://closure-af.dzhk.de/